CLINICAL TRIAL: NCT07065032
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Multiple-ascending-dose Phase Id/IIa Study Evaluating the Safety, Tolerability, and Pharmacokinetics of ZT002 Injection in Adult Chinese Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Study of ZT002 Injection in Adult Chinese Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJQLZT002DM003
Record Dates: First submitted 2025-06-06; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZT002 Injection dose 1 (Experimental): Dose 1 administered subcutaneously, Q2W
  Interventions: Drug: ZT002 Injection
- ZT002 Injection dose 2 (Experimental): Dose 2 administered subcutaneously, Q2W
  Interventions: Drug: ZT002 Injection
- ZT002 Placebo (Placebo Comparator): Placebo administered subcutaneously, Q2W
  Interventions: Drug: ZT002 Placebo

INTERVENTIONS:
Drug: ZT002 Injection — Q2W, subcutaneous injection
  Arms: ZT002 Injection dose 1
Drug: ZT002 Injection — Q2W, subcutaneous injection
  Arms: ZT002 Injection dose 2
Drug: ZT002 Placebo — Participants will receive the same volume as the study drug in each cohort.
  Arms: ZT002 Placebo

SUMMARY:
This study will comprise a randomized, double blind, placebo controlled, multiple ascending dose, safety, tolerability and pharmacokinetic study of ZT002 in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blind, placebo-controlled, multiple-ascending-dose Phase Id/IIa clinical study in Chinese T2DM subjects after diet and exercise intervention and/or treatment with oral hypoglycemic agent to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical efficacy of ZT002 injection in adult subjects with type 2 diabetes mellitus. Participants in each cohort will be randomized to receive a multiple SC doses of either ZT002 or matching placebo every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 65 years (inclusive, based on age at the time of signing the informed consent form);
2. Body mass index (BMI) at screening ranges from 22-35 kg/m² (inclusive); BMI = Weight(kg)/ Height (m²).
3. Type 2 diabetes mellitus has been diagnosed for ≥12 weeks according to the diagnostic and classification criteria for diabetes mellitus issued by the World Health Organization (WHO) in 1999 and the WHO Recommendations for Diagnosis Using Glycosylated Hemoglobin (HbA1c) (2011) supplemental diagnostic criteria; and one of the following conditions is met:

   1. Controlled by diet and exercise for 12 weeks prior to screening, with no prior use of any hypoglycemic drugs
   2. Use of only one oral hypoglycemic agent (including metformin, α-glucosidase inhibitors, dipeptidyl peptidase-4 [DPP-4] inhibitors, and sodium-glucose cotransporter 2 [SGLT2] inhibitors) in the 12 weeks prior to screening, but no further use in the 14 days prior to screening;
4. At screening and before randomization: 7.0% ≤ glycosylated hemoglobin (HbA1c) ≤ 10.5% (hospital laboratory);
5. At screening and before randomization: fasting venous blood glucose ≤ 13.9 mmol/L (hospital laboratory);

Exclusion criteria (Subjects meeting any of the following criteria will not be enrolled in the trial):

1. History of specific allergies (asthma, eczema, etc.) or allergic constitution, or history of allergy to two or more drugs and foods, especially to the investigational drug and its excipients or GLP-1-containing drugs;
2. Confirmed or suspected diagnosis of type 1 diabetes mellitus or specific types of diabetes mellitus (monogenic diabetes syndrome, cystic fibrosis, pancreatitis, drug or chemically induced diabetes mellitus, etc.) for other causes prior to screening;
3. History of acute and chronic pancreatitis, history of symptomatic gallbladder disease (except for cholecystectomy), history of pancreatic injury, and other high risk factors for pancreatitis prior to screening;
4. Previous personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia syndrome (MEN2); or hyperthyroidism or hypothyroidism on stable dose medication for less than 3 months;
5. Diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic syndrome (HHS), diabetic lactic acidosis, or hyperosmolar nonketotic diabetic coma within 12 months prior to screening;
6. Proliferative retinopathy, maculopathy, symptomatic diabetic neuropathy, intermittent claudication, and diabetic foot that are unstable or require treatment within 12 months prior to screening;
7. Severe hypoglycemic (grade 3 hypoglycemic) events within 6 months prior to screening, or 3 or more hypoglycemic events (blood glucose < 3.9 mmol/L) within 1 month prior to randomization, or recurrent hypoglycemia-related symptoms (1 or more per week) prior to randomization;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events and serious adverse events; Number of participants with injection site reaction. | up to 155days

SECONDARY OUTCOMES:
Area under the concentration-time curve at the end of dosing interval(τ) at steady state (AUC0-τ,SS) | up to 155days
Time to Cmax at steady state (Tmax,ss) | up to 155days
Steady-state peak concentration (Css_max), mean steady-state concentration (Css_av) | up to 155days
Change from baseline of venous fasting plasma glucose | up to 155days
Change from baseline of weight (kg). | up to 155days
Incidence of anti-drug antibody against ZT002 | up to 155days

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, PhD, Principal Investigator — The Affiliated Hospital of Qingdao University; Chengqian Li, MD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No